CLINICAL TRIAL: NCT05120063
Title: Benefit of 3-D Planning in Total Hip Replacement. A Prospective Randomized Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Collaborators: Symbios Orthopedie SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: KEK Nr. 2012-0064
Record Dates: First submitted 2021-05-06; First posted 2021-11-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Hip Injuries; Surgery; Prosthesis User
MeSH Terms: conditions — Hip Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 3D anatomical stem (Experimental): 3-D-Planing with anatomical stem (SPS monoblock stem, Symbios)
  Interventions: Device: SPS monoblock stem, Symbios; Procedure: 3D planning of THR
- 3D non-anatomical stem (Experimental): 3-D-Planing with non anatomical stem (Quadra-H, Medacta)
  Interventions: Device: Quadra-H, Medacta; Procedure: 3D planning of THR
- 2D anatomical stem (Experimental): 2-D-Planing with anatomical stem (SPS monoblock stem, Symbios)
  Interventions: Device: SPS monoblock stem, Symbios; Procedure: 2D planning of THR
- 2D non anatomical stem (Experimental): 2-D-Planning with non anatomical Stem (Quadra-H, Medacta)
  Interventions: Device: Quadra-H, Medacta; Procedure: 2D planning of THR

INTERVENTIONS:
Device: SPS monoblock stem, Symbios — hip prosthesis
  Arms: 2D anatomical stem; 3D anatomical stem
Device: Quadra-H, Medacta — hip prosthesis
  Arms: 2D non anatomical stem; 3D non-anatomical stem
Procedure: 3D planning of THR — primary total-hip replacement (THR) planned on 3-dimensional images (computer tomography)
  Arms: 3D anatomical stem; 3D non-anatomical stem
Procedure: 2D planning of THR — primary total-hip replacement (THR) planned on 2-dimensional images (anteroposteiros pelciv x-ray)
  Arms: 2D anatomical stem; 2D non anatomical stem

SUMMARY:
In this prospective randomized four-armed study the investigators aim to compare wheter 3-D planning, which necessitates preoperative CT acquisition and sophisticated planning together with engineers, results in measurable benefits in terms of objective and subjective outcome values in a collective of patients undergoing primary total hip replacement.

Hypothesis:

1. When compared to 2-D planning, 3-D planning of a THR results in better hip reconstruction, better subjective and clinical outcome and better longevity of total hip implants.
2. When compared to a non-anatomical stem, an anatomical stem allows better hip reconstruction, better subjective and clinical outcome and better longevity of total hip implants.

DETAILED DESCRIPTION:
Patients sent to our outpatient clinic for eventual primary THR are informed about this study and written patient information given to them. When patients decide to undergo primary total hip replacement, patient's questions with respect to this study are discussed in the outpatient clinic and patients willing to participate included.

Block randomization using closed envelopes for age categories 40-50, 50-60, 60-70 years will be conducted to assign the participant to one of the four study arms.

Patients will be blinded for the type of stem and method of planning. Investigators are blined in terms of methods of planning. In terms of stem design, investigators can not be blinded since their visibility on x-ray does not allow it.

The preoperative investigation includes routine investigation and an additional CT scan plus evaluation of the "University of California at Los Angeles" (UCLA) activity level and "Short Form Health 36" (SF-36) score. The same applies for the postoperative investigation and 3 months. The follow-up visits at 1, 5 and 10 years are routine investigations with additional UCLA and SF-36 Scores.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 40-70 years scheduled for primary THR
* signed written informed consent.

Exclusion Criteria:

* Charnley class B and C
* ASA score >2
* pregnancy
* gross hip deformity making complex hip reconstruction (greater trochanter advancement, acetabular augmentation, femoral osteotomy, use of cemented or revision stem) necessary
* immature patients and patients incompetent to judge

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2030-01-28 (Estimated); Study Completion 2030-01-28 (Estimated)

PRIMARY OUTCOMES:
Change in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Change from basline to one year
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients, including pain, stiffness, and physical functioning of the hip.
  A difference in WOMAC of 2.5 points is considered relevant. 3-D-planing and/or anatomical stems will be considered superior to 2-D-planing and /or non-anatomical stems if the one year WOMAC significantly differs by 2.5.
Change in subjective hip value (SHV) | Change from basline to one year
  The subjective hip value (SHV) is as a patient-reported outcome measurement (PROM) which is reported by the patient. It is easily and quickly performed and interpreted. The SHV is defined as a patient's subjective hip satisfaction expressed as a percentage of 100%, which is the score that an entirely normal hip joint would reach.
  A difference in subj. hip value of 25% is considered relevant. 3-D-planing and/or anatomical stems will be considered superior to 2-D-planing and /or non-anatomical stems if the one year subjective hip value significantly differs by 25%.